CLINICAL TRIAL: NCT02753686
Title: Treatment of Canadian Men and Pre/Postmenopausal Women With ER+ Advanced Breast Cancer in the Real-World Setting With Hormone Therapy ± Targeted Therapy
Brief Title: Treatment of Canadian Men and Pre/Peri/Post-menopausal Women With ER+ Advanced Breast Cancer in the Real-World Setting With Hormone Therapy ± Targeted Therapy
Acronym: Treat ER+ight
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRAD001YCA09
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: HR+ HER2- Men, Pre/Postmenopausal Advanced Breast Cancer
Keywords: HR+ HER2; pre/postmenopausal; men; advanced breast cancer; non steroidal aromatase inhibitor (NSAI) exposure; metastatic; endocrine therapy; targeted therapy; prospective; observational; registry; real world setting; adult; CRAD001; non-interventional; Canadian; CDK; cyclin dependent kinase
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Neoplasm Metastasis | interventions — Anastrozole; exemestane; Tamoxifen; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Endocrine Therapy (ET): HR+ HER2- male, female pre/postmenopausal advanced breast cancer patients being treated with endocrine therapy
  Interventions: Drug: Endocrine therapy may include one of the following therapies: letrozole, anastrozole, exemestane, tamoxifen or fulvestrant
- Cohort 2: Endocrine Therapy (ET) plus Targeted Therapy (TT): HR+ HER2- male, female pre/ postmenopausal advanced breast cancer patients being treated with endocrine therapy in combination with targeted therapy including CDK4/6 inhibitor therapy
  Interventions: Drug: Endocrine therapy in combination with targeted therapy may include: everolimus plus exemestane or CDK4/6 inhibitor plus endocrine therapy

INTERVENTIONS:
Drug: Endocrine therapy may include one of the following therapies: letrozole, anastrozole, exemestane, tamoxifen or fulvestrant
  Groups: Cohort 1: Endocrine Therapy (ET)
Drug: Endocrine therapy in combination with targeted therapy may include: everolimus plus exemestane or CDK4/6 inhibitor plus endocrine therapy
  Groups: Cohort 2: Endocrine Therapy (ET) plus Targeted Therapy (TT)

SUMMARY:
Although randomized controlled trials (RCTs) provide evidence of efficacy, generalization of these results to patients in the real-world setting is challenging, given RCTs are conducted in highly selected patient populations.

An understanding of the effectiveness of approved cancer therapies in routine clinical practice is essential in order to optimize the management of these patients and to identify treatment and monitoring gaps.

This is the first Canadian study to describe real-world treatment patterns/sequencing, effectiveness and monitoring for men and pre/postmenopausal HR+ HER2- advanced breast cancer patients. This registry incorporates an observational prospective cohort design and will enroll 500 men and pre/postmenopausal HR+ HER2- advanced breast cancer women that have been exposed to endocrine therapy (ET) or ET in combination with targeted therapy (TT) including patients receiving CDK4/6 inhibitor therapy combinations..

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient is an adult, male or female ≥ 18 years old at the time of informed consent.
2. Patient has histologically and/or cytologically confirmed diagnosis of breast cancer.
3. Patient has inoperable locally advanced or metastatic breast cancer.
4. Patient has ER positive and/or PgR positive HER2-negative breast cancer by local laboratory testing (based on most recently analyzed biopsy).
5. In the case of women, both pre/perimenopausal and postmenopausal patients are allowed to be included in this study.

   1. Postmenopausal status is defined as per investigator's judgment. Definition included as guidance only:

1. Prior bilateral oophorectomy 2. Or age ≥60 3. Or age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifen, or ovarian suppression), and FSH and estradiol in the postmenopausal range per local normal range. If patient is taking tamoxifen or toremifene and age < 60, then FSH and plasma estradiol levels should be in postmenopausal range per local normal range.

b) Premenopausal status is defined as per investigator's judgment. Definition included as guidance only:

1. Patient had last menstrual period within the last 12 months 2. Or if on tamoxifen or toremifene within the past 14 days, plasma estradiol and FSH must be in the premenopausal range per local normal range 3. Or in case of therapy induced amenorrhea, plasma estradiol and/or FSH must be in the premenopausal range per local normal range.

c) Perimenopausal status is defined as neither premenopausal nor postmenopausal as per investigator's judgment.

6. Patient having received maximum one prior chemotherapy line for advanced/metastatic breast cancer is allowed.

Note: A chemotherapy line in advanced disease is an anticancer regimen(s) that contains at least 1 cytotoxic chemotherapy agent and given for 21 days or longer. If a cytotoxic chemotherapy regimen was discontinued for a reason other than disease progression and lasted less than 21 days, then this regimen does not count as a "prior line of chemotherapy".

7. Patient receiving targeted therapy plus endocrine therapy (ET+TT) in either the 1st, 2nd or 3rd line or endocrine therapy alone (ET) in either the 2nd or 3rd line advanced metastatic setting:

1. as per approved Health Canada indication OR
2. as per available expanded treatment protocol(s) only if efficacy assessments in these protocols are considered routine standard of care OR
3. as per available compassionate / expanded access program

   Notes: 1. Date of initiation of treatment should be a maximum of 12 months prior to the date of enrollment in this study for patients receiving CDK4/6 inhibitor therapy based combinations. Date of initiation of treatment should be a maximum of 1 month prior to the date of enrollment in this study for patients receiving all other endocrine monotherapies or combination therapies. 2. 1st, 2nd and 3rd line therapy in the advanced setting is defined as the first, second and third treatment received respectively in the metastatic setting (which could include endocrine monotherapy, targeted therapy combination with endocrine therapy or chemotherapy). 3. 3. Patients enrolled in the ET cohort must have received a prior CDK4/6 inhibitor for advanced/metastatic breast cancer. Patients who have received two subsequent lines of CDK4/6 inhibitor therapy are allowed.

   8. The decision to use ET or ET+TT has been reached prior to and independently of the current study.

   9. Patient willing to be followed according to routine standard of care practice.

   10. Signed informed consent to allow the collection of the data for the purposes of this study.

   EXCLUSION CRITERIA:
   1. Patient currently receiving chemotherapy at baseline/study entry is excluded (however patient could have received up to one line of chemotherapy in the metastatic setting prior to study entry or as a subsequent therapy after completion of ET or ET+TT treatment).
   2. Patient having received more than 3 lines of therapy in the metastatic setting.
   3. Any contraindications to the study treatments as presented in the respective Canadian Product Monographs for each therapy.
   4. Patient is participating in a clinical trial for an investigational treatment with the exception expanded treatment protocol or access program where efficacy assessments are considered routine standard of care.
   5. Patient is undergoing any treatment that is not considered standard of care as per regional policies and guidelines with the exception of treatments accessed via expanded treatment protocols or access programs.
   6. Patient does not understand or is not willing to sign the informed consent for participation in the study.
   7. According to the judgment of the physician participation in the study may interfere with the treatment or compromise the well-being of the patient.
   8. Patient is expected to travel for an extensive time period or be unavailable during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian men, pre/postmenopausal women with advanced HR+ HER2- breast cancer and currently receiving endocrine therapy (ET) or ET plus targeted therapy (TT).
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Duration on Treatment | Up to approximately 24 months
  To describe the duration on treatment with ET and ET+TT by cohort subgroups defined by (but not limited to) previous treatment with a CDK4/6 inhibitor plus endocrine therapy combination and according to the current line of treatment for advanced breast cancer up to and including 3rd line

SECONDARY OUTCOMES:
Treatment Sequencing | Up to approximately 72 months
  To describe the sequence of therapies and treatment patterns used for the management of advanced breast cancer.
Monitoring Patterns | Up to approximately 72 months
  To characterize monitoring patterns associated with complete blood count (CBC), liver function tests (LFT), electrolytes and electrocardiogram (ECG) specifically in patients treated with CDK4/6-based combinations.
Overall Survival (OS) | Up to approximately 72 months
  To describe the therapeutic effectiveness of endocrine therapy (ET) and ET in combination with targeted therapy (TT) as measured by OS.
Health Care Resource Utilization (HCRU) | Up to approximately 72 months
  To describe HCRU related to management of advanced breast cancer.
Health Related Quality of Life (HRQoL - EORTC QLQ-C30) | Up to approximately 72 months
  To describe the change in HRQoL EORTC 30 questionnaire QLQ-C30
HRQoL BR23 | Up to approximately 72 months
  To describe the change in HRQoL Breast Cancer 23 Questionnaire BR23
Work-Related Productivity | Up to approximately 72 months
  To describe the change in work-related productivity.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- Canada (20):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, North Vancouver, British Columbia
  - Novartis Investigative Site, Richmond, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Sault Ste. Marie, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
  - Novartis Investigative Site, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doyle C, Lohmann AE, Iqbal N, Henning JW, Kulkarni S, Califaretti N, Hilton J, Ferrario C, Bouganim N, Mates M, Guillemette S, Leite R, Caron MA, Thireau F, Machado A, Chia S. A Canadian real-world, multi-center, prospective, observational study assessing the treatment duration, the treatment sequence, and the overall survival for patients treated with endocrine therapy +/- targeted therapy in HR + HER2-negative advanced breast cancer. Breast Cancer Res Treat. 2025 Apr;210(2):425-438. doi: 10.1007/s10549-024-07580-8. Epub 2025 Jan 23. PMID 39847203